CLINICAL TRIAL: NCT02811692
Title: CODEX:Collection of Aflibercept Data in Routine Practice
Brief Title: Study for Collection of Aflibercept Data in Routine Practice
Acronym: CODEX
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 17867; DBOX 2014/00498 (Other: Company Internal)
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Eye Diseases
Keywords: Database; Diabetic Macular Edema (DME); Wet Age-related Macular Degeneration (wAMD); Retinal Diseases; Optic Nerve Diseases; Corneal Diseases; Vision Disorders
MeSH Terms: conditions — Eye Diseases; Retinal Diseases; Optic Nerve Diseases; Corneal Diseases; Vision Disorders | interventions — aflibercept

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- BAY86-5321: Anti-Vascular Endothelial Growth Factor (VEGF) - naive patients starting intravitreal Aflibercept injection treatment for Neovascular age-related macular degeneration (AMD), macular edema following Branch Retinal Vein Occlusion (BRVO), macular edema following central retinal vein occlusion (CRVO), and diabetic macular edema (DME)
  Interventions: Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321) — Administration by intravitreal injection

SUMMARY:
The French CODEX study is designed as a national database to describe, in routine medical practice, functional and anatomical responses to intravitreal Aflibercept injection, in a large population of anti-VGEF-naïve patients presenting with wet Age-related Macular Degeneration (wAMD), Central Retinal Vein Occlusion (CRVO),Branch Retinal Vein Occlusion(BRVO), or Diabetic Macular Edema (DME). This national database will gather databases from French private and public ophthalmologic centers.

DETAILED DESCRIPTION:
The retrospective data will be gathered from the first injection of Aflibercept for the indications macular edema following Branch Retinal Vein Occlusion (BRVO) directly by each physician. For each patient, the first injection date of Aflibercept is defined as the index date.

Electronic files from each ophthalmologist, containing patient medical records, will be periodically transmitted according to the milestones of the study with a maximum of 4 transfers (at Q2 2016 for the first transfer and then every 9 months thereafter).

As each electronic transfer will be independent of each other and as patients' data will be anonymized by physicians before each transfer, data comparisons will be not possible between the four electronic files transfers planned over the study period.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years old
* Anti-VEGF (Vascular Endothelial Growth Factor) treatment naïve
* Intravitreal (IVT) aflibercept injection treatment follows the recommendations made within the EYLEA Summary of Product Characteristics
* Diagnosed with wAMD (wet Age-related Macular Degeneration), macular edema following CRVO (Central Retinal Vein Occlusion), macular edema following BRVO (Branch Retinal Vein Occlusion), or DME (Diabetic Macular Edema).

Exclusion Criteria:

* Who have any contraindications listed in the EYLEA Summary of Product characteristics
* Participating in an investigational program with interventions outside of routine clinical practice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult naïve patients (not previously treated with an anti-VEGF agent) with diagnosis of wet Age-related Macular Degeneration (wAMD), macular edema following Branch Retinal Vein Occlusion (BRVO), macular edema following central retinal vein occlusion (CRVO), and Diabetic Macular Edema (DME) and starting treatment with Aflibercept.
Sampling Method: Non-Probability Sample
Enrollment: 425 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2017-11-27 (Actual)

PRIMARY OUTCOMES:
Change in Best Corrected Visual Acuity (BCVA) using Early Treatment Diabetic Retinopathy Study (ETDRS) or converted to ETDRS. | Baseline and 12 months
Change in Central retinal thickness (CRT) as measured by Optical Coherence Tomography (OCT). | Baseline and 12 months

SECONDARY OUTCOMES:
Change in Best Corrected Visual Acuity (BCVA) using Early Treatment Diabetic Retinopathy Study (ETDRS) or converted to ETDRS. | Baseline and 6 month, 18 month and 24 month
  in each indication
Change in Central retinal thickness (CRT) as measured by Optical Coherence Tomography (OCT). | Baseline and 6 month, 18 month and 24 month
  in each indication
Number of injections | Baseline and 6 month, 12 month, 18 month and 24 months
  in each indication
Interval (days) between injections per disease | Baseline and 6 month, 12 month, 18 month and 24 months
  in each indication
Presence of pigment epithelial detachment (PED) (Y/N) | Baseline and 6 month, 12 month, 18 month and 24 months
  In wet age-related macular degeneration (wAMD) population
Proportion of patients with no fluid determined by OCT (absence of fluid includes all types of fluid and location of fluid as determined by the treating ophthalmologist) | Baseline and 6 month, 12 month, 18 month and 24 months
Type of adjunctive therapies (ie focal laser, steroids etc.) | Baseline and 6 month, 12 month, 18 month and 24 months
Change in score of diabetic retinopathy as determined by treating ophthalmologist | Baseline and 6 month, 12 month, 18 month and 24 months
  In Diabetic Macular Edema (DME) population

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, France